CLINICAL TRIAL: NCT06683209
Title: Comparison of Scleral Indentation Instruments and Impact on Patient Comfort
Brief Title: Optimizing Patient's Comfort During Scleral Indentation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of Toronto (Other); Alberta Retina Consultant (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00146504
Record Dates: First submitted 2024-10-31; First posted 2024-11-12 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Pain
Keywords: Schocket; Josephberg-Besser; Cotton tip applicator
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: In each group, patient receive two different types of scleral depressor, one in each eye.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): One eye examined with the Schocket scleral depressor, the other eye with the Josephberg-Besser scleral depressor
  Interventions: Diagnostic Test: Schocket scleral depressor; Diagnostic Test: Josephberg-Besser
- Group B (Active Comparator): One eye examined with the Schocket scleral depressor, the other eye with the cotton tip applicator
  Interventions: Diagnostic Test: Schocket scleral depressor; Diagnostic Test: Cotton tip applicator
- Group C (Active Comparator): One eye examined with the cotton tip applicator, the other eye with the Josephberg-Besser scleral depressor
  Interventions: Diagnostic Test: Josephberg-Besser; Diagnostic Test: Cotton tip applicator

INTERVENTIONS:
Diagnostic Test: Schocket scleral depressor — Use of this instrument to examine one eye
  Arms: Group A; Group B
Diagnostic Test: Josephberg-Besser — Use of this instrument to examine one eye
  Arms: Group A; Group C
Diagnostic Test: Cotton tip applicator — Use of this instrument to examine one eye
  Arms: Group B; Group C

SUMMARY:
The scleral depression exam is an important routine technique for evaluating the retinal periphery for various reasons. During this examination, an instrument is used to bring the anterior part of the retina into the physician's field of view. The downside of this technique is the discomfort it may cause the patient. Different instruments can be used to depress the sclera.

The objective of this research is to compare three commonly used scleral depressors based on their performance for the ophthalmologist and the discomfort they subjectively induce in patients.

Patients will be randomly allocated to one of three examination groups:

Group A: One eye examined with the Schocket scleral depressor, the other eye with the Josephberg-Besser scleral depressor.

Group B: One eye examined with the Schocket scleral depressor, the other eye with the cotton-tip applicator.

Group C: One eye examined with the cotton-tip applicator, the other eye with the Josephberg-Besser scleral depressor.

DETAILED DESCRIPTION:
Background The scleral depression exam is an important technique for evaluating the retinal periphery during indirect ophthalmoscopy. Despite the advent of ultra-widefield fundus imaging, scleral depression provides greater sensitivity in detecting peripheral lesions, such as retinal tears. It was found that 11% of retinal tears were missed when employing non-contact slit-lamp examination, compared to indirect ophthalmoscopy with scleral depression, and a scleral depression exam is widely considered the gold standard for ruling out retinal tears. While there is no international consensus, the preferred practice guideline (American Academy of Ophthalmology) for assessing peripheral vitreoretinal pathology is by indirect ophthalmoscopy combined with scleral depression.

There are a variety of ophthalmic instruments that an eye care professional may use to perform scleral depression. While the exam is uncomfortable, there is a lack of studies comparing patient comfort with different instruments. In this prospective study, we will compare subjective patient pain scores using the Schocket scleral depressor, the Josephberg-Besser scleral depressor, and the cotton-tipped applicator.

Purpose To assess patient pain scores for three common scleral indentation devices and determine which is most comfortable for patients.

Objective / Hypothesis Based on clinical experience, the hypothesis is that the Josephberg-Besser scleral depressor causes less discomfort due to its design.

Study Design Prospective comparative analysis.

Methods Patients will be recruited at two tertiary referral centers (Alberta Retinal Consultants, Edmonton, Alberta, and Sunnybrook Hospital, Department of Ophthalmology & Vision Sciences, Toronto, Ontario) upon consent to participate. Subject identification will be based on the referral indication (symptomatic posterior vitreous detachment with or without vitreoretinal pathology) and the absence of exclusion criteria (i.e., patients who require a scleral indentation examination based on the presenting symptoms). Patients will then be randomly allocated to one of three groups. Additionally, within each group, the symptomatic eye will be randomized.

Patients will be dilated with 1% tropicamide and 2.5% phenylephrine for 30 minutes. Instillation of local anesthetic drops will be used to eliminate any confounding exposure-related keratalgia or ocular surface irritation. Indirect ophthalmoscopic evaluation of the retinal periphery will be undertaken using the provider's lens of choice (20 or 28-diopter lens). The lens and illumination settings will be kept the same for each eye. A similar amount of time and effort will be spent on both eyes.

Following the examination, both patients and physicians will be asked to provide responses to the survey questions provided (surveys enclosed).

Statistical analysis will be performed using R statistical software. Randomization to treatment will be created using Python programming software.

Exclusions:

Monocular status. Media opacity that precludes view of the peripheral retina. Inadequate examination (cooperation with examination, inability to achieve all directions of gaze).

Underlying oculodynia (recent surgery, intraocular inflammation, abnormal intraocular pressure, ocular dysesthesia syndromes (ocular, adnexal, or orbital)).

History of pain-sensitizing conditions or current analgesic use. Previous scleral indentation examination poorly tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic posterior vitreous detachment with or without vitreoretinal pathology

Exclusion Criteria:

* Monocular status.
* Media opacity which precludes view of the peripheral retina.
* Inadequate examination (cooperation with examination, inability to achieve all directions of gaze).
* Underlying oculodynia (recent surgery, intraocular inflammation, abnormal intraocular pressure, ocular dysesthesia syndromes (ocular, adnexal or orbital).
* History of pain-sensitizing conditions or current analgesic use.
* Previous scleral indented examination poorly tolerated.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Pain scale | Once, directly after completing the scleral depressed examination, on the same day of inclusion in the study.
  Patient rate their pain with the Wong-Baker Faces scale for each eye, from 0 to 10, 0 being the absence of pain and 10 being the worst imaginable pain.

SECONDARY OUTCOMES:
Ergonomics Ease of use | Once, directly after completing the scleral depressed examination, on the same day of inclusion in the study.
  Physician rate their proficiency with the scleral depressor used
  o No difficulty o Some difficulty o Significant difficulty
Performance accessing the visualized area | Once, directly after completing the scleral depressed examination, on the same day of inclusion in the study.
  Physician rate their proficiency with the scleral depressor used
  o No difficulty o Some difficulty o Significant difficulty
Quantity of indentation | Once, directly after completing the scleral depressed examination, on the same day of inclusion in the study.
  Physician rate their proficiency with the scleral depressor used. Indentation area of the medium light setting of the ophthalmoscope while using a 28D lens. Small is less than 1/3, medium is between 1/3 and 2/3, large is more than 2/3.
Performance achieving sufficient indentation | Once, directly after completing the scleral depressed examination, on the same day of inclusion in the study.
  Physician rate their proficiency with the scleral depressor used
  o No difficulty o Some difficulty o Significant difficulty
Duration of examination | Time mesure will be during the examination of each eye
  The scleral depressed examination will be timed to ensure a similar duration between each eye
Degree of retinal pathology | The physician will note his findings right after his examination, while completing his examination survey
  The physician will annotate his findings based on the number and the type of retinal pathology (tear, hole, lattice, other) found.

OTHER OUTCOMES:
Depressor routinely used by participating physician | Before recruiting patients
  Participating physician must state their routine instrument for scleral depression.
  o Schocket o Josephberg-Besser o Cotton tip applicator
Lens routinely used by participating physician | Before recruiting patients
  Participating physician must state their routinely used lens for scleral depression 20 diopters or 28 diopters

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Alberta Retina Consultant, Edmonton, Alberta
  - Sunnybrook Hospital, Toronto, Ontario